CLINICAL TRIAL: NCT02865265
Title: Association Between Ultrasound-guided Pecs II Block and Parasternal Block May Represent a Valid Alternative for the Management of Acute and Postoperative Pain Syndrome in Breast Cancer Surgery: a Retrospective Study
Brief Title: Pecs II Block and PaB Could be an Alternative in Breast Surgery
Status: Completed | Type: Observational
Sponsor: Emiliano Petrucci (Other)
Responsible Party: Sponsor-Investigator, Emiliano Petrucci, Dr Emiliano Petrucci, San Salvatore Hospital of L'Aquila
Organization: San Salvatore Hospital of L'Aquila (Other)
Other Study IDs: 0109060/16
Record Dates: First submitted 2016-08-04; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pecs II and parasternal blocks: Pecs II block was performed at the level of the fourth rib in the fascial plane between the minor pectoral and serratus anterior muscles, and 20 ml of 0.5% levobupivacaine solution were injected.
  An ultrasound-guided ipsilateral PaB was performed via two separate injections of 4 ml of 0.375% levobupivacaine at the level of the 2nd and 4th intercostal space underneath the external intercostal membrane between the major pectoral and intercostal muscles close to the surface of the 2nd and 4th rib.
  Interventions: Procedure: Pecs II and parasternal blocks

INTERVENTIONS:
Procedure: Pecs II and parasternal blocks — Pecs II block was performed at the level of the fourth rib in the fascial plane between the minor pectoral and serratus anterior muscles, and 20 ml of 0.5% levobupivacaine solution were injected.
  An ultrasound-guided ipsilateral parasternal block was performed via two separate injections of 4 ml of 0.375% levobupivacaine at the level of the 2nd and 4th intercostal space underneath the external intercostal membrane between the major pectoral and intercostal muscles close to the surface of the 2nd and 4th rib.

SUMMARY:
The association between ultrasound-guided Pecs II block and parasternal block can represent a valid alternative in the management of acute and postoperative pain syndrome after quadrantectomy with or without axillary dissection.

DETAILED DESCRIPTION:
The combination of Pecs II block and PaB provides good management of postoperative pain and can be considered a viable alternative to common anesthetic procedures performed for breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age;
* American Society of Anesthesiologists (ASA) physical status I-III,
* patients scheduled for quadrantectomy with or without axillary dissection

Exclusion Criteria:

* pregnancy;
* body mass index (BMI) >35;
* allergy to local anesthetics;
* skeletal or muscle abnormalities of the chest wall;
* presence of primary or secondary neurological diseases;
* presence of psychiatric diseases;
* history of chronic pain or neuropathic disorders;
* history of drug abuse;
* state of sepsis;
* infection
* tumors of the skin on the chest;
* primary;
* secondary coagulopathies

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for quadrantectomy with or without axillary dissection.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2013-03; Primary Completion 2013-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pain | Pain was recorded at 24 months after surgery
  Pain has been evaluate with visual analogue scale (VAS) at 24 months after surgery

SECONDARY OUTCOMES:
Neuropathic postoperative disturbances | Neuropathic postoperative disturbances were recorded at 24 months after surgery
  Neuropathic postoperative disturbances were examined using the von Frey hair test (neuropathic disturbances: present/not present) at 24 months
Patient satisfaction | Patient satisfaction was evaluated at 1 day after surgery
  Patient satisfaction with regard to the anesthetic procedure was assessed using a five-step satisfaction scale (not at all/slightly/somewhat/very/extremely satisfied).
Woud healing | Wound healing was assessed at 24 months after surgery
  Wound healing was assessed using a three-step scale (unacceptable/acceptable/excellent healing) in accordance with the surgeon's opinion.

IPD SHARING:
Plan to Share IPD: No